CLINICAL TRIAL: NCT06583928
Title: Frequency of Refeeding Syndrome in Critically Ill Children At Assiut University Hospital
Brief Title: Refeeding Syndrome in Critically Ill Children
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Manal Mohamed Ali, Principal investigator, Assiut University
Other Study IDs: Refeeding syndrome Frequency
Record Dates: First submitted 2024-08-31; First posted 2024-09-04 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Refeeding Syndrome; Syndrome, Refeeding
MeSH Terms: conditions — Refeeding Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Refeeding syndrome (RFS) is the a metabolic disturbance which occurs as a result of reinstitution of nutrition in people who are starved, severely malnourished, or metabolically stressed because of severe illness. When too much food or liquid nutrition supplement is eaten during the initial three to seven days following a malnutrition event, the production of glycogen, fat and protein in cells may cause low serum concentrations of potassium, magnesium and phosphate.

DETAILED DESCRIPTION:
Refeeding syndrome (RFS) is the a metabolic disturbance which occurs as a result of reinstitution of nutrition in people who are starved, severely malnourished, or metabolically stressed because of severe illness. When too much food or liquid nutrition supplement is eaten during the initial three to seven days following a malnutrition event, the production of glycogen, fat and protein in cells may cause low serum concentrations of potassium, magnesium and phosphate.

When risk factors are not identified and nutrition therapy is not managed appropriately, devastating consequences such as electrolyte depletion and imbalances, fluid overload, arrhythmia, seizure, encephalopathy, and death may occur.

Once nutrition is reintroduced to a patient who has been starved for an extended period, anabolism begins directly . The body shifts back to carbohydrate metabolism from protein and fat catabolism, and glucose becomes the primary source of energy once again. The increased glucose load, with a corresponding increase in the release of insulin, leads to cellular uptake of glucose, potassium, magnesium,and phosphate. This shift of electrolytes back into the cell causes,hypokalemia,hypomagnesemia, and hypophosphatemia. Insulin also exhibits a natriuretic effect on the kidneys. Hence, sodium is retained, causing fluid retention and expansion of the extracellular fluid volume.

Hypophosphatemia is the hallmark of RFS. Other electrolyte abnormalities are associated with RFS, however, such as hypokalemia and hypomagnesemia. Shifts in glucose, sodium, and fluid balance are also seen in RFS. Consequently, cardiovascular, pulmonary, neuromuscular, hematologic, and gastrointestinal complications occur.

This syndrome can emerge with aggressive oral nutrition, enteral nutrition, or PN and can be fatal if not recognized and treated in a timely manner.

Refeeding syndrome can be fatal if not recognized and treated properly. The electrolyte disturbances of the refeeding syndrome can occur within the first few days of refeeding. Close monitoring of blood biochemistry is therefore necessary in the early refeeding period.

A Data on RFS incidence is lacking, and the heterogeneity of diagnostic criteria and frequent electrolyte disorders in this population make its diagnosis complex. In 2020, the American Society for Parenteral and Enteral Nutrition (ASPEN) developed consensus recommendations for identifying patients at risk and with refeeding syndrome. These state that undernourished children are considered at risk of refeeding syndrome; those who develop one significant electrolyte disorder (decrease ≥ 10% in phosphorus, potassium, and/or magnesium) within the first five days of nutritional support, combined with a significant increase in energy intake, are considered to have refeeding syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Children included were those (1month to 18 years) admitted at hospital with minimum of one phosphorus, potassium, and/or magnesium assay and who are severely malnourished and starved (no feeding )for at least 3 days then received exclusive or supplemental nutritional support.

Undernourished children (body mass index z-score < -2 standard deviations) were considered at risk of refeeding syndrome. The ASPEN critiera were used to identify those with probable refeeding syndrome.

Exclusion Criteria:

* Patients age less than 1month and more than 18 years' old and patients with CKD ,liver cirrhosis and endocrinal diseases.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: - Children (1month to 18 years) admitted at hospital with minimum of one phosphorus, potassium, and/or magnesium assay and who are severely malnourished and starved (no feeding )for at least 3 days then received exclusive or supplemental nutritional support.
  Undernourished children (body mass index z-score < -2 standard deviations) were considered at risk of refeeding syndrome. The ASPEN critiera were used to identify those with probable refeeding syndrome.
Sampling Method: Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Determine the numbers of patients who developed refeeding syndrome according to ASPEN criteria , those who develop one significant electrolyte disorder (decrease ≥ 10% in phosphorus, potassium, and/or magnesium) within the first | Basline

REFERENCES:
- [Background] Runde J, Sentongo T. Refeeding Syndrome. Pediatr Ann. 2019 Nov 1;48(11):e448-e454. doi: 10.3928/19382359-20191017-02. PMID 31710364
- [Background] Doig GS, Simpson F, Heighes PT, Bellomo R, Chesher D, Caterson ID, Reade MC, Harrigan PW; Refeeding Syndrome Trial Investigators Group. Restricted versus continued standard caloric intake during the management of refeeding syndrome in critically ill adults: a randomised, parallel-group, multicentre, single-blind controlled trial. Lancet Respir Med. 2015 Dec;3(12):943-52. doi: 10.1016/S2213-2600(15)00418-X. Epub 2015 Nov 18. PMID 26597128
- [Background] Mehanna HM, Moledina J, Travis J. Refeeding syndrome: what it is, and how to prevent and treat it. BMJ. 2008 Jun 28;336(7659):1495-8. doi: 10.1136/bmj.a301. No abstract available. PMID 18583681
- See also: Related Info — https://scholar.google.com/scholar?hl=en&as_sdt=0%2C5&pq=refeeding+syndrome+in+children&oq=#d=gs_qabs&t=1721590022186&u=%23p%3DEZjkMYnXzD0J
- See also: Related Info — https://doi.org/10.3389/fped.2022.932290
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC9253668/